CLINICAL TRIAL: NCT01599039
Title: Prospective Controlled Study Comparing the Effectiveness and Specificity of Inverse Water Volumetry Versus Bio-impedance Spectroscopy in the Assessment of Early Recognition of Breast Cancer Related Lymphoedema.
Brief Title: Study the Usefulness of Bio-impedance Spectroscopy in the Early Assessment of Breast Cancer Related Lymphoedema
Status: Completed | Type: Observational
Sponsor: Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, R.J. Damstra, Dermatologist MD PhD, Nij Smellinghe Hosptial
Other Study IDs: NS3NL
Record Dates: First submitted 2012-05-13; First posted 2012-05-15 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Lymphedema; Breast Cancer Stage II; Early Disease Onset
Keywords: early diagnostics; lymphedema; breast cancer; breast cancer related lymphedema; measuring methods; inverse water volumetry; prevention
MeSH Terms: conditions — Lymphedema; Breast Neoplasms; Breast Cancer Lymphedema

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- breast cancer patients with SN: 1. Breast cancer patients with sentinel node biopsy (n=25)
- breast cancer patients with AD: 2. Breast cancer patients with axillary dissection (n=25)
- colo-rectal patients: 3. Colo-rectal patients as control group (n=25)

SUMMARY:
The goal of the study is to investigate the use of bio-impedance spectroscopy in the assessment of breast cancer related lymphoedema in patients operated with lumpectomy or mastectomy, axillary lymph node dissection and radiotherapy compared to inverse water volumetry. As a control group, patients with colon rectal cancer are used to compare volumetric and spectometric changes during follow-up.

DETAILED DESCRIPTION:
Current assessment of lymphoedema consists of measuring volume changes objectively by a tape measure or water displacement. Early recognition of pre-clinical changes of interstitial fluid congestion in a limb at risk concerning lymph transport capacity is crucial. Objective measurement of extracellular fluids with bio-impedance spectroscopy can detect these early signs of lymphoedema. Multi Frequency Bioelectrical Impedance Analysis is completely non-invasive, highly reproducible (Ward et al 1997), highly sensitive (Cornish et al 2001), highly specific (Cornish et al 2001) and can be repeated as frequently as desired. BIS demonstrated excellent inter- and intra-rater reliability. All measures are highly reliably in women with and without lymphoedema (Szerniec et al 2010). For women with lymphoedema BIS detected a difference in the ECF in limbs which were not reflected in a corresponding difference in limb volume. This finding suggests that BIS may be particularly useful in the early detection of lymphoedema, before there is any volume change (Szerniez et al 2010). The mean ratio of extra cellular water (ECW) to intracellular water (ICW) is 1,5:1 (Ward et al 2009). Cornish et al (2001) predicted the onset of the condition up to 10 months before the condition could be clinically diagnosed. This is considerable shorter than the mean delay time of 3,5 years reported by National Summit on Lymphoedema, Adelaide 2000. The only risk factor identified as contributing to an increased risk of developing secondary lymphoedema was an increasing BMI which is consistent with previous reports (Box et al 2002).

Early detection with BIS is supposed possible even before clinical signs of swelling are available.

In this study we want to study this hypothesis and as control-group patients treated for colorectal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Gender: female
* Patients operated with lumpectomy or mastectomy, Sentinel node, axillary lymphnode dissection and/or chemotherapy and/or radiotherapy.
* Controls: operated for colon-rectal carcinoma with colectomy and adjuvant chemotherapy
* Patients 18 years or older
* No pre-existing clinical or volumetric signs of lymphoedema (CBO guideline: >10% difference with contra-lateral side

Exclusion Criteria:

* Allergy against one of the used materials
* Patients who have a pacemaker or other inbuilt stimulator
* Women who are pregnant
* Patients with renal failure or heart failure
* Lymphoedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There study population consists of breast cancer patients treated with either sentinel node biopsy either axillary dissection. As a control group we use colorectal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Bio impedance spectometry | 2 years
  The participant's height (to 1 mm) and weight (to 0.1 kg) are measured prior to BIS assessment and entered into the device for processing. Whole arm impedance (wrist to axilla) will be determined according to the principle of equipotentials; a method shown to have greater precision than a 'paired electrode' approach. Participants were positioned in supine on a non-conductive bed with their arms by their side, pronated and slightly abducted. These result are compared with the gold standard (Inverse watter volumetry)

SECONDARY OUTCOMES:
body Mass Index (BMI) | 2 years
  The body mass index (or BMI) is a measure which shows whether people have the right weight for their height. The World Health Organisation (WHO), governments and health workers use it. It is also called the Quetelet Index.
quality of life measurement with the " LAST" meter | 2 years
  The "lastmeter" is a validated tool in the Dutch language to score the psycho-social and physical situation of a cancer patient. The scale is between 0-10 and includes several questions. This indicates the need for addition support by healthcare workers to improve QoL

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Damstra, PhD, Principal Investigator — Nij smellinghe hospital, Netherlands
Locations (1):
- Expert Center for Lymphovascular Medicine Nij Smellinghe Hospital, Drachten, Provincie Friesland, Netherlands

REFERENCES:
- See also: The foundation related to the expert centre organizing research — http://www.slcn.nl
- See also: General website form the Nij Smellinghe hospital — http://www.nijsmellinghe.nl